CLINICAL TRIAL: NCT03532412
Title: Different Loop Gain Phenotypes in Patients With Chronic Systolic Heart Failure and Periodic Breathing
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_LoopGain
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Periodic Breathing
Keywords: Polysomnography, Sleep apnea, Central sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HF+CSA+PB: Systolic heart failure with predominant central sleep apnea and periodic breathing

SUMMARY:
Central sleep apnoea (CSA) is common in patients with chronic systolic heart failure (HFrEF). Various trials have shown a prevalence of 21 - 37% in this group of people. Up to 66% of patients with CSA and HFrEF present with periodic breathing (PB), which is considered being a marker of HF severity and poor prognosis. Brack et al. summarized data from cohorts, longitudinal studies and retrospective analyses showing an independently increased risk of death in HF patients with PB (HR 2.1-5.7 in five of seven studies). Furthermore, PB in HF patients is known to reduce quality of life and exercise performance and to increase sympathetic nerve activity as well as the probability of malignant cardiac arrhythmias.

The pathogenesis of PB is characterized by an instability of ventilatory drive. The level of carbon dioxide (CO2) in blood and cerebrospinal fluid correlates linearly with minute ventilation. A high level of CO2 increases ventilation while hypocapnia dampens it. This control theory is based on the loop gain (LG), which represents the sensitivity and reactivity of the ventilatory system and comprises three components: The plant gain defines the capacity of the system to change PaCO2 in response to a change in ventilation (metabolic response). It is influenced by the lung volume as well as the anatomy of the thorax and the upper airways. The feedback gain is defined by the chemoreceptor responsiveness in reaction to blood gas changes. The controller gain is represented by the respiratory control center in the brain stem and defines the capacity of the system to change ventilation in response to a change in PaCO2 (ventilatory response).

Sands et al. proposed and validated a mathematical model based on the ventilatory cycle pattern that quantifies the feedback loop. The ratio of ventilatory and cycle duration within the PB pattern is defined as the duty ratio (DR), which is the basis to calculate the LG. Any temporary breathing disturbance causing a PB pattern with a LG < 1 stabilizes within a few breathing cycles. A LG > 1 represents an unstable ventilatory response and slight changes of CO2 are accompanied by overshooting and undershooting of the ventilation. In that case, the polysomnography shows the typical pattern of waxing and waning of the tidal volume and effort.

HF patients typically present with an increased LG due to an impaired left ventricular function and a hyperstimulation of pulmonary vagal receptors. Furthermore, Khoo showed an increased chemosensitivity (controller gain) as well as a decreased ventilatory capacity (plant gain) in this group of people.

Sands and colleagues characterized PB considering the mean LG derived from several ventilatory cycles during non-REM sleep. This retrospective study of PB in HFrEF patients addresses the following questions:

1. Is a single LG value appropriate to characterize the individual PB?
2. Does the LG depend on sleep stage and body position?
3. Does the intraindividual LG variability allow for the discrimination of different PB phenotypes and, if so, do these phenotypes differ in further characteristics?

ELIGIBILITY:
Inclusion Criteria:

* Systolic heart failure with left-ventricular ejection fraction <45%
* Apnea-Hypopnea index >15 per hour as determined by diagnostic polysomnography
* Predominant central sleep apnea as defined by >50% central respiratory events

Exclusion Criteria:

* <50 evaluable respiratory events for loop gain analysis during diagnostic polysomnography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the sleep lab for diagnostic polysomnography.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Loop Gain | During one day of diagnostic polysomnography
  Mathematically determined loop gain of periodic breathing according to Sands et al. [10] based on diagnostic polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Director
Locations (1):
- Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brack T, Randerath W, Bloch KE. Cheyne-Stokes respiration in patients with heart failure: prevalence, causes, consequences and treatments. Respiration. 2012;83(2):165-76. doi: 10.1159/000331457. Epub 2011 Oct 18. PMID 22025128
- [Background] Javaheri S, Shukla R, Zeigler H, Wexler L. Central sleep apnea, right ventricular dysfunction, and low diastolic blood pressure are predictors of mortality in systolic heart failure. J Am Coll Cardiol. 2007 May 22;49(20):2028-34. doi: 10.1016/j.jacc.2007.01.084. Epub 2007 May 4. PMID 17512359
- [Background] Naughton MT. Epidemiology of central sleep apnoea in heart failure. Int J Cardiol. 2016 Mar;206 Suppl:S4-7. doi: 10.1016/j.ijcard.2016.02.125. Epub 2016 Feb 26. PMID 26948168
- [Background] Randerath W, Verbraecken J, Andreas S, Arzt M, Bloch KE, Brack T, Buyse B, De Backer W, Eckert DJ, Grote L, Hagmeyer L, Hedner J, Jennum P, La Rovere MT, Miltz C, McNicholas WT, Montserrat J, Naughton M, Pepin JL, Pevernagie D, Sanner B, Testelmans D, Tonia T, Vrijsen B, Wijkstra P, Levy P. Definition, discrimination, diagnosis and treatment of central breathing disturbances during sleep. Eur Respir J. 2017 Jan 18;49(1):1600959. doi: 10.1183/13993003.00959-2016. Print 2017 Jan. PMID 27920092
- [Background] Yumino D, Bradley TD. Central sleep apnea and Cheyne-Stokes respiration. Proc Am Thorac Soc. 2008 Feb 15;5(2):226-36. doi: 10.1513/pats.200708-129MG. PMID 18250216
- [Background] Kasai T, Floras JS, Bradley TD. Sleep apnea and cardiovascular disease: a bidirectional relationship. Circulation. 2012 Sep 18;126(12):1495-510. doi: 10.1161/CIRCULATIONAHA.111.070813. No abstract available. PMID 22988046
- [Background] Rowley JA, Badr MS. Central Sleep Apnea in Patients with Congestive Heart Failure. Sleep Med Clin. 2017 Jun;12(2):221-227. doi: 10.1016/j.jsmc.2017.03.001. PMID 28477776
- [Background] Naughton MT. Loop gain in apnea: gaining control or controlling the gain? Am J Respir Crit Care Med. 2010 Jan 15;181(2):103-5. doi: 10.1164/rccm.200909-1449ED. No abstract available. PMID 20053968
- [Background] Wellman A, Malhotra A, Fogel RB, Edwards JK, Schory K, White DP. Respiratory system loop gain in normal men and women measured with proportional-assist ventilation. J Appl Physiol (1985). 2003 Jan;94(1):205-12. doi: 10.1152/japplphysiol.00585.2002. Epub 2002 Sep 20. PMID 12391042
- [Background] Sands SA, Edwards BA, Kee K, Turton A, Skuza EM, Roebuck T, O'Driscoll DM, Hamilton GS, Naughton MT, Berger PJ. Loop gain as a means to predict a positive airway pressure suppression of Cheyne-Stokes respiration in patients with heart failure. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1067-75. doi: 10.1164/rccm.201103-0577OC. PMID 21816941
- [Background] Khoo VS. MRI--"magic radiotherapy imaging" for treatment planning? Br J Radiol. 2000 Mar;73(867):229-33. doi: 10.1259/bjr.73.867.10817036. No abstract available.